CLINICAL TRIAL: NCT06472206
Title: Community Health Workers And MHealth to ImProve Viral Suppression Plus (CHAMPS+)
Acronym: CHAMPS+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Alabama at Birmingham (Other); Health Services Center, Inc. (Unknown); Unity Wellness Center (Unknown); Louisiana State University Health Sciences Center in New Orleans (Other); University of Mississippi Medical Center (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Tulane University (Other)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Professor of Disease Prevention and Health Promotion and Professor of Population and Family Health; Associate Dean of Faculty Development, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAU8885; R01MD019184 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): The control condition includes standard health services offered at each site. All participants receive referrals to mental health, drug/alcohol treatment, and/or other HIV services as necessary. Standard of care at each site follows the Dept. of Health and Human Services HIV guidelines.
- Intervention CHAMPS+ (Experimental): Participants randomized to intervention will receive the CleverCap pill bottle, an innovative technology that dispenses only the prescribed amount of medication, keeps track of medications dispensed, and communicates wirelessly with the WiseApp. Additionally, participants will receive 10-12 sessions with CHWs, and sexual health log to keep track of their sexual behavior.
  Interventions: Behavioral: CHW Sessions; Device: CleverCap

INTERVENTIONS:
Behavioral: CHW Sessions — Sessions with a Community Health Worker (CHW).
  Arms: Intervention CHAMPS+
Device: CleverCap — The CleverCap pill bottle is an innovative technology that dispenses only the prescribed amount of medication, keeps track of medications dispensed, and communicates wirelessly with the WiseApp to deliver medication adherence reminders.
  Arms: Intervention CHAMPS+

SUMMARY:
Although global efforts have been made to end the HIV epidemic, there are still some gaps in HIV testing, antiretroviral therapy (ART) adherence, and viral suppression (VS) among people with HIV (PWH). These gaps are particularly prominent in the Deep South of the United States (US), where PWH face challenges in accessing healthcare services. In response, a team of experienced researchers has developed and tested the Community Health Workers And MHealth to ImProve Viral Suppression (CHAMPS) intervention. This intervention uses mobile health (mHealth) technology and a team of community health workers (CHW) to design an intervention to improve ART adherence and VS. The CHAMPS+ intervention adds a CHW delivered supportive risk reduction counseling during periods of non-suppression to prevent HIV transmission. The study will engage the participants by developing culturally relevant materials and retention strategies, evaluating the clinical effectiveness and sustainability of the intervention in Deep South settings, and assessing regionalized implementation factors. Ultimately, the study will test the effectiveness of CHAMPS+ on ART adherence and viral load suppression for PWH in Alabama, Louisiana, and Mississippi.

DETAILED DESCRIPTION:
Despite efforts to achieve UNAIDS 95-95-95 targets, marked deficits remain in HIV testing, antiretroviral therapy (ART) adherence, and viral suppression (VS) among a growing number of persons with HIV (PWH). Gaps in HIV treatment success are particularly pronounced in the United States (US) Deep South. These suboptimal HIV health outcomes occur at a time when clinicians have limited time and the US healthcare system remains fragmented, further exacerbating the challenges inherent in the lives of underserved, marginalized groups, such as PWH. In this way, the development and evaluation of interventions using a resource-savvy cadre of community health workers (CHW) holds promise for addressing these challenges. Yet, gaps exist in the CHW literature, and research is needed to bring CHW interventions to scale to ameliorate the large gaps in the US HIV Care Continuum, particularly in Ending the HIV Epidemic (EHE) priority locations.

In response, the study team has developed and tested the Community Health Workers And MHealth to ImProve Viral Suppression (CHAMPS) intervention which leverages mobile health (mHealth) technology to create a multi-component intervention that targets multiple levels (individual, social and sexual networks, and community) to improve ART adherence and VS. The study team will build on the strong preliminary data of extant intervention work in PWH by leveraging the CHAMPS intervention which will be delivered by personnel from four HIV care settings in the Deep South. The CHAMPS+ intervention is delivered via an mHealth platform to support PWH to self-manage their ART regimens and adds to the extant CHAMPS intervention by adding a CHW-delivered supportive risk reduction counseling (sexual behavior and substance use) during periods of non-suppression to prevent HIV transmission. This study also builds upon mChoice (U01PS005229) and WiseApp (R01HS025071) studies to improve ART adherence and VS in the Deep South. This study design has a three-fold purpose of: 1) engaging the target population in the development of culturally relevant recruitment materials and retention strategies for the study, 2) assessing the clinical effectiveness and sustainability of the intervention in Deep South settings, and 3) evaluating regionalized implementation factors guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance framework. Ultimately, this study will test CHAMPS+ to promote ART adherence and suppressed viral load for PWH in in Alabama, Louisiana (Orleans Parish), and Mississippi, US EHE prioritized jurisdictions. Importantly, the multi-component intervention targets multiple levels to address HIV risk behaviors during periods of non-suppression--an innovative and impactful component likely to be of great public health import.

ELIGIBILITY:
Inclusion Criteria:

* Be able to speak, read, and write in English;
* Be above 18 years of age;
* Be willing to participate in any assigned arm of the intervention;
* Have an HIV-1 RNA level >200 copies/mL;
* Own a smartphone;
* Be able and willing to provide informed consent for study participation and consent for access to medical records.
* Live, work and or receive care in AL, LA, or MS

Exclusion Criteria:

* Reside in a nursing home, prison, and/or receiving in-patient psychiatric care at time of enrollment;
* Terminal illness with life expectancy <6 months; and
* Planning to move out of the area in the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2027-07-22 (Estimated); Study Completion 2027-12-22 (Estimated)

PRIMARY OUTCOMES:
Change in Viral Load | Baseline, 6 month follow up, 12 month follow up.
  Using blood samples obtained during standard of care visits, viral load levels will be used to asses ART adherence.

SECONDARY OUTCOMES:
Change in ART adherence - CleverCap. | Up to 12 months.
  The CleverCapTM dispenser will automatically record each time a participant opens the dispenser. The investigators will collect adherence data from participants in the intervention arm each day from the start to the end of trial (day 1 to 12 months), and it is a count response (number of times taking medication each day).
Change in Score on the Self-Rating Scale Item (SRSI). | Baseline, 6 month follow up, 12 month follow up.
  The Self-Rating Scale Item is a single-item self-report adherence measure that uses a 5-point Likert scale to describe medication adherence over the past 4 weeks. The total score range is 1(very poor) to 6 (excellent). A higher score indicates higher self-reported adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, Principal Investigator — Columbia University; Scott Batey, PhD, MSW, Principal Investigator — Tulane University
Locations (5):
- United States (5):
  - Health Services Center, Inc., Hobson City, Alabama
  - Unity Wellness Center, Opelika, Alabama
  - Louisiana State University Health Sciences Center in New Orleans, New Orleans, Louisiana
  - Tulane University, New Orleans, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi